CLINICAL TRIAL: NCT05386069
Title: The Effect of a Non-Opioid Multimodal Pain (NOMO) Protocol in Decreasing Narcotic Use After Urogynecologic Surgery
Brief Title: Does a Non-Opioid Multimodal Pain (NOMO) Protocol Decrease Narcotic Use
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NOMO Protocol
Record Dates: First submitted 2020-04-06; First posted 2022-05-23 (Actual); Results first posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Opioid Use
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Arm (No Intervention): Routine Care per Anesthiologist/cRNA
- Treatment Arm (Active Comparator): Patients to receive standard weight-based ketamine bolus (0.5 mg/kg) at start of procedure, withhold opioids in post-operative period unless rescue medications fail
  Interventions: Drug: NOMO Protocol

INTERVENTIONS:
Drug: NOMO Protocol — Standard weight-based ketamine bolus (0.5 mg/kg) at procedure start, no Opioid rescue medications
  Other Names: Standard Care
  Arms: Treatment Arm

SUMMARY:
The objective of this study is to evaluate narcotic use after implementation of a Non-Opioid Multimodal Pain (NOMO) protocol in patients who are undergoing a urogynecologic procedure. The study will also evaluate secondary outcomes, including: post-operative pain rating, length of hospital stay, postoperative antiemetic use, bladder catheterization at discharge, number of post-operative phone calls, and rate of reported side effects of opioid use (nausea/constipation). Study participants will be asked to utilize the validated Brief Pain Inventory (appendix A) scale to assess post-operative pain levels. Based on inpatient post-operative opioid use and number of opioid pills prescribed at discharge, an attempt will be made to develop an algorithm for recommended opioid prescribing patterns.

DETAILED DESCRIPTION:
The objective of this study is to evaluate narcotic use after implementation of a Non-Opioid Multimodal Pain (NOMO) protocol in patients who are undergoing a urogynecologic procedure. NOMO protocols seek to reduce the opioid usage for patients in the postoperative period. Patients will receive multiple pain medications (usually referred to as a "pain cocktail") that work on various pain receptors throughout the body. These medications are approved for pain control; but they have few side effects and less addictive properties. The study will also evaluate secondary outcomes, including: post-operative pain rating, length of hospital stay, postoperative antiemetic use, bladder catheterization at discharge, number of post-operative phone calls, and rate of reported side effects of opioid use (nausea/constipation). Study participants will be asked to utilize the validated Brief Pain Inventory (appendix A) scale to assess post-operative pain levels. Based on inpatient post-operative opioid use and number of opioid pills prescribed at discharge, an attempt will be made to develop an algorithm for recommended opioid prescribing patterns.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking females
* greater than or equal to 18 years old
* scheduled for a urogynecologic procedure at GHS requiring inpatient stay or extended observation.

Exclusion Criteria:

* less than 18 years of age
* non-English speaking patients
* unscheduled urogynecologic surgeries
* patients expected to undergo a simple reconstructive surgery with same-day discharge,
* history of chronic pain
* chronic Lyrica or Celebrex use
* psychiatric disorder, narcotic dependence or narcotic prescription in the past six weeks
* current liver disease
* kidney disease (defined as GFR <60)
* malignancy
* sulfa allergy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Females undergoing Urogynecology procedure
Enrollment: 10 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hema Brazell, MD, Principal Investigator — Prisma Health
Locations (1):
- Prisma Health - Upstate, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Reagan KML, O'Sullivan DM, Gannon R, Steinberg AC. Decreasing postoperative narcotics in reconstructive pelvic surgery: a randomized controlled trial. Am J Obstet Gynecol. 2017 Sep;217(3):325.e1-325.e10. doi: 10.1016/j.ajog.2017.05.041. Epub 2017 May 25. PMID 28551445

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Arm | Treatment Arm
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | Treatment Arm | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10
Brief Pain Inventory (Short Form) [Median (Full Range); unit: units on a scale] | 4.8 [1 to 10] | 2.4 [1 to 10] | 3.6 [1 to 10]

OUTCOME MEASURES:

1. Primary Outcome: Morphine Milligram Equivalents Used During Inpatient Stay
Description: Total morphine milligram equivalents calculated for each patient during their stay.
Time Frame: from immediately postoperative through discharge or 4 weeks, whichever comes first
Population: Patients undergoing urogynecologic procedure.
Measure: Mean (Standard Deviation); unit: morhpine milligram equivalents
Arm/Group | Control Arm | Treatment Arm
Number analyzed (Participants) | 5 | 5
morhpine milligram equivalents | 10.8 (5.6) | 8.8 (7.1)

2. Secondary Outcome: Passage of Voiding Trial
Description: percentage of patients who pass voiding trial on POD#1
Time Frame: from immediately postoperative through discharge or 4 weeks, whichever comes first
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Treatment Arm
Number analyzed (Participants) | 5 | 5
Participants | 4 | 4

3. Secondary Outcome: Anti-emetic Use
Description: Did the patient require anti-emetics in the post-operative period
Time Frame: postoperative day 1 through day of discharge from hospital; all patients were dischard on post-op day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Treatment Arm
Number analyzed (Participants) | 5 | 5
Participants | 5 | 5

4. Secondary Outcome: Patient Pain Score
Description: Evaluated via the "Brief Pain Inventory (Short Form)"; rate pain on scale 0-10, 10 being worst
Time Frame: postoperative day 7
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Control Arm | Treatment Arm
Number analyzed (Participants) | 5 | 5
score on a scale | 4.8 [0 to 10] | 2.4 [0 to 10]

5. Secondary Outcome: Prescription for Opioid at Discharge
Description: Did the patient require a narcotic prescription
Time Frame: postoperative day 2 through postoperative day 7
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Treatment Arm
Number analyzed (Participants) | 5 | 5
Participants | 4 | 1

6. Secondary Outcome: Length of Hospital Stay
Description: The average number of days patients were admitted as inpatient.
Time Frame: postoperative day 1 through discharge or 4 weeks, whichever comes first
Population: All enrolled patients included - all patients stayed in hospital for 2 days.
Measure: Mean (Full Range); unit: days
Arm/Group | Control Arm | Treatment Arm
Number analyzed (Participants) | 5 | 5
days | 2 [2 to 2] | 2 [2 to 2]

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Control Arm | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-21): https://cdn.clinicaltrials.gov/large-docs/69/NCT05386069/Prot_SAP_000.pdf